CLINICAL TRIAL: NCT03990324
Title: Immediate Changes in Cervical Range of Motion and Myofascial Sensitivity After Standardized Manual Stretches: a Randomized Controlled Trial
Brief Title: Cervical Range of Motion and Stretching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: University of Indianapolis (Other); Nova Southeastern University (Other); Long Island University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIO-17-13405
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Cervical Shortening
Keywords: range of motion; muscle sensitivity; muscle stretching

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessor of dependent variables was blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group did not received intervention and sat on a table for approximately 5 minutes
- Stretching group (Experimental): The stretching group received a standardized manual stretching protocol
  Interventions: Procedure: Manual stretching

INTERVENTIONS:
Procedure: Manual stretching — Manual stretching for the upper trapezius and levator scapulae muscle
  Arms: Stretching group

SUMMARY:
Cervical range of motion (ROM) is necessary to perform normal activities of daily living and deficits are associate with various pathologies. Currently, its unclear if specific myofascial stretches will improve cervical range of motion and decrease myofascial sensitivity. After a single session of the manual stretching procedure, participants immediately demonstrated increased cervical ROM and pressure pain thresholds.

DETAILED DESCRIPTION:
Methods: Sixty participants with no history of neck pain or trauma were randomized into one of two groups: stretching group (n = 30), or control group (n = 30). The stretching group received a standardized manual stretching protocol. The control group did not received intervention. Pre and Post-test measurements were recorded for both groups. Within group differences and group by time interactions were evaluated for Cervical range of motion ROM and myofascial sensitivity. The immediate improvement in active ROM of the cervical spine may prompt clinicians to consider the sequencing of treatment. Stretching prior to active exercises may allow for active exercise through a larger ROM. Future research is needed to evaluate the immediate effects of stretching in the symptomatic population.

ELIGIBILITY:
Inclusion Criteria:

* ages of 18-60
* active cervical flexion, right lateral flexion OR left cervical lateral flexion <45˚

Exclusion Criteria:

* minors
* prisoners
* individuals with cognitive impairments
* recent neck surgeries
* pre-existing neck injuries

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Range of Motion | 1 minute post-intervention
  CROM including flexion, extension, side bending left, side bending right, rotation left, and rotation right

SECONDARY OUTCOMES:
Pressure pain thresholds | 1 minute post-intervention
  The PPT was recorded using a Wagner FDX-25 hand-held digital pressure algometer (Wagner Instruments, Greenwich, CT). The investigator performed each assessment uniformly by applying force at the same rate of 5 Pa/second.

CONTACTS AND LOCATIONS:
Overall Officials: William J Hanney, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No